CLINICAL TRIAL: NCT03668795
Title: Surgical Management of Placenta Accreta a Three Year Experience at King Hussein Medical Center
Brief Title: Surgical Management of Placenta Accreta
Status: Completed | Type: Observational
Sponsor: Royal Medical Services, Jordanian Armed Forces (Other)
Responsible Party: Principal Investigator, Mitri Rashed, Dr. Mitri Rashed, senior specialist in obstetrics and gynaecology and IVF, Royal Medical Services, Jordanian Armed Forces
Other Study IDs: RoyalMSJordan
Record Dates: First submitted 2018-09-11; First posted 2018-09-13 (Actual); Last update posted 2018-09-17 (Actual); Status verified 2018-09

CONDITIONS: To Publish Our Experience in the Surgical Management to Placenta Accreta Cases and the Maternal Outcome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Bakrey balloon insertion within the uterus and caesarean hysterectomy — Creating an intrauterine tamponade to stop the uterine bleeding by inflating an intrauterine balloon with 600 cc of saline versus undergoing hysterectomy if conservative management failed
  Other Names: Interventional radiological insertion of balloon to obstuct the internal iliac artery

SUMMARY:
purpose of this study was to report our experience for surgical management of suspected placenta accreta cases encountered in King Hussein medical center

DETAILED DESCRIPTION:
was a retrospective study of all patients who underwent planned deliveries for placenta accreta at King Hussein Medical Centre (KHMC) from August 2011 to October 2014.Demographic characteristics were recorded. Ultrasound (U/S) and magnetic resonance imaging (MRI) were used for the diagnosis. Surgery for all patients were performed by multidisciplinary teams. All information were obtained from patient's files.

ELIGIBILITY:
Inclusion Criteria:

* all placenta previa accreta cases encountered in our institution over three year period

Exclusion Criteria:

-

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All pregnant ladies who were diagnosed to have placenta previa accreta cases which was diagnosed using ultrasound or MRI
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2011-08-01 (Actual); Primary Completion 2014-10-30 (Actual); Study Completion 2017-11-30 (Actual)

PRIMARY OUTCOMES:
The intraoperative and short term postoperative complications of surgical interventions in placenta accreta | 48 hours
  Intraoperative visceral injuries, bleeding, and short term postoperative morbidity and mortality

IPD SHARING:
Plan to Share IPD: Undecided